CLINICAL TRIAL: NCT05873556
Title: Development and Preliminary Examination of Two Brief Personalized Feedback Interventions Focused on Lab-based and EMA Alcohol Cues to Reduce Hazardous Young Adult Alcohol Use
Brief Title: Testing Brief Personalized Feedback Integrating Lab-based Alcohol Cue Information
Acronym: Project ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jason Ramirez, Acting Assistant Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016989; R34AA027302 (NIH)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions: (1) Personalized feedback based on reports from baseline and lab-session and (2) assessment-only control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lab-based Cue Reactivity Personalized Feedback Intervention (PFI) (Experimental): Participants randomized to the Lab-based Cue Reactivity PFI condition view the online personalized feedback in the lab after completing the cue reactivity protocol. Participants view the feedback on their own during the lab session. The personalized feedback is delivered online and contains information summarizing participants' desire to drink, mood, willingness to drink, and alcohol demand as reported before and after alcohol exposure.
  Interventions: Behavioral: Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
- Assessment-only control (No Intervention): Participants randomized to the control group do not receive any intervention. They complete all the survey assessments and the lab-based cue reactivity protocol without ever receiving any personalized feedback.

INTERVENTIONS:
Behavioral: Lab-based Cue Reactivity Personalized Feedback Intervention (PFI) — This is an online personalized feedback intervention that contains information summarizing participants' desire to drink, mood, willingness to drink, and alcohol demand as reported before and after alcohol exposure.
  Arms: Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)

SUMMARY:
This study aims to develop a brief intervention that uses information from a lab-based cue reactivity protocol to create personalized feedback targeting high-risk alcohol use among young adults who drink alcohol. The intervention provides feedback on individuals' drinking desire, mood, willingness to drink, and alcohol demand by comparing scores before and after viewing and smelling an alcoholic beverage in the lab session. Other psycho-educational alcohol-related content is also provided in the intervention including strategies for decreasing exposure to cues that increase drinking desires and how to cope with increased desire to drink. This brief intervention is used in a randomized controlled trial (RCT) comparing young adults who receive the brief, online intervention to those who did not receive the brief, online intervention. Participants in both groups complete baseline, lab-based cue reactivity protocol, 2-week follow-up and 3-month follow-up.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test a brief intervention that provides personalized feedback to young adults using participants' responses from a baseline survey and from a lab-based cue reactivity protocol. The aim of the intervention is to increase young adults' awareness of how alcohol cues may affect their desire to drink, mood, willingness to drink, and alcohol demand both in relation to lab-based exposure to an alcohol beverage of their choice and also more broadly in everyday life. The intervention also aims to equip young adults with strategies for reducing exposure to factors that increase their desire to drink, how to cope with an increased desire to drink, and how to reduce potential harms from drinking.

This brief personalized feedback intervention is used in a randomized controlled trial comparing young adults who receive the intervention with those who complete the assessments and lab protocol but do not receive any personalized feedback. Online assessments include an eligibility survey, baseline assessment, and follow-up assessments occurring 2-weeks and 3-months post-intervention. Everyone has one in-person session to complete the lab-based cue reactivity protocol after the baseline assessment has been completed online. The intervention will be examined for its feasibility, acceptability, and its effects in reducing alcohol-related outcomes at the follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-24
* Lives in Washington state
* Reports drinking at least two days per week in the last six months
* Reports at least one heavy drinking episode (4+/5+ drinks for women/men) in the past month
* Open to changing drinking behavior
* Must be willing to come to our Seattle study office for session visit
* Provide an email address and phone number for study communication

Exclusion Criteria:

* Actively seeking treatment for alcohol use
* Currently participating in another study in our research center regarding young adult drinking behavior

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ramirez, PhD, Principal Investigator — University of Washington; Anne Fairlie, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share limited, de-identified datasets for the purposes of data analysis and dissemination.
Time Frame: Data dictionaries and limited datasets can be made available starting in May 2024.
Access Criteria: Individual requests to access data with intended purpose should be made to Drs. Fairlie and Ramirez and will be reviewed by the investigative team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Washington state (e.g., via Instagram). Individuals were invited to complete an online eligibility survey for participation in a randomized clinical trial to test the effect of an online personalized feedback intervention. Recruitment (i.e., posting ads on social media) went from April 2023 to December 2023. Participant enrollment (i.e., completion of lab session) went from May 2023 to December 2023.
Groups:
- Assessment-only Control: Participants randomized to the control group will not receive any intervention. They complete all the survey assessments and the lab-based cue reactivity protocol without ever receiving any personalized feedback.
- Lab-based Cue Reactivity Personalized Feedback Intervention (PFI): Participants randomized to the Lab-based Cue Reactivity PFI condition will receive a link to the personalized feedback in the lab after completing the cue reactivity protocol. Participants view the feedback on their own during the lab session. The personalized feedback is delivered online and contains information summarizing participants' desire to drink, mood, willingness to drink, and alcohol demand as reported before and after alcohol exposure.
  Lab-based Cue Reactivity Personalized Feedback Intervention (PFI): This is an online personalized feedback intervention that contains information summarizing participants' desire to drink, mood, willingness to drink, and alcohol demand as reported before and after alcohol exposure.
Period: Overall Study
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
Started | 42 | 51
Completed | 38 | 50
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI) | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 51 | 93
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.93 (1.66) | 21.04 (1.87) | 21.44 (1.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 36 | 42 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 26 | 35 | 61
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 51 | 93
Student Status [Count of Participants; unit: Participants]
  4-year student | 21 | 30 | 51
  Not a 4-year student | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Daily Drinking Questionnaire
Description: Number of standard drinks consumed on each day of a typical week during the [past 3 months for baseline and 3-month follow-up; past two weeks for 2-week follow-up]. Participants responded on a scale from 0 (0 drinks) to 25 (25 or more drinks). Totals for each day are summed to calculate the typical number of drinks consumed per week.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Measure: Mean (Standard Deviation); unit: Drinks per week
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 42 | 51
Drinks per week
  Baseline | 10.24 (5.16) | 12.27 (7.95)
  2-Week Follow-Up | 8.79 (7.25) | 9.73 (6.95)
  3-Month Follow-Up | 6.97 (5.46) | 9.14 (7.70)
Statistical Analysis 1: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=93 with a Condition × 2-Week Follow-Up interaction. AOC was the reference category for Condition, and Baseline was the reference category for 2-Week Follow-Up; p = 0.83, Generalized linear mixed model; Models controlled for sex assigned at birth, age, and student status (4-year vs. not) and used a Poisson error distribution; Count/Rate Ratio = 0.97, 95% CI 2-sided [0.74 to 1.27]
Statistical Analysis 2: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=93 with a Condition × 3-Month Follow-Up interaction. AOC was the reference category for Condition, and Baseline was the reference category for 3-Month Follow-Up; p = 0.61, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.07, 95% CI 2-sided [0.83 to 1.38]

2. Primary Outcome: Heavy Episodic Drinking
Description: Participants were asked, "During the past two weeks, how many times did you have [4/5 for females/males] or more drinks at one sitting?". Participants responded on a scale from 0 (0 times) to 10 (10 or more times) and possible range was 0-10.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Measure: Mean (Standard Deviation); unit: Heavy Drinking Occasions
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 42 | 51
Heavy Drinking Occasions
  Baseline | 2.45 (1.92) | 2.47 (2.17)
  2-Week Follow-Up | 1.86 (1.78) | 2.18 (1.75)
  3-Month Follow-Up | 1.53 (1.37) | 1.86 (1.95)
Statistical Analysis 1: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.45, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.16, 95% CI 2-sided [0.79 to 1.72]
Statistical Analysis 2: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.46, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.17, 95% CI 2-sided [0.77 to 1.79]

3. Primary Outcome: Penn Alcohol Craving Scale
Description: Self-reported subjective alcohol craving during the past week. Response options were scored from "0" to "6" with text varying across items. A sum score of the five items was calculated and the possible range was from 0-30. Higher scores reflect more craving.
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 42 | 51
Score on a scale
  Baseline | 6.93 (3.96) | 8.04 (4.11)
  2-Week Follow-Up | 7.31 (4.81) | 8.04 (5.44)
  3-Month Follow-Up | 5.74 (4.23) | 7.24 (5.09)
Statistical Analysis 1: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.62, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 0.95, 95% CI 2-sided [0.77 to 1.17]
Statistical Analysis 2: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.34, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.14, 95% CI 2-sided [0.87 to 1.48]

4. Primary Outcome: Brief Young Adult Alcohol Consequences Questionnaire
Description: Participants responded "no" (0) or "yes" (1) to whether they experienced each of 24 consequences during the [past 3 months for baseline and 3-month follow-up; past two weeks for 2-week follow-up]. A sum of the number of negative alcohol-related consequences was calculated and the possible range was 0-24. Higher values represent a worse outcome (i.e., more consequences).
Time Frame: Baseline, 2 week follow-up, and 3 month follow-up
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
Number analyzed (Participants) | 42 | 51
Score on a scale
  Baseline | 8.74 (5.18) | 9.92 (5.02)
  2-Week Follow-Up | 4.88 (4.80) | 5.78 (5.11)
  3-Month Follow-Up | 6.11 (5.26) | 7.06 (5.37)
Statistical Analysis 1: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 2-Week Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.66, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.08, 95% CI 2-sided [0.76 to 1.54]
Statistical Analysis 2: Comparison: Assessment-only Control vs Lab-based Cue Reactivity Personalized Feedback Intervention (PFI); Changes from Baseline to 3-Month Follow-Up for PFI versus AOC reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.92, Generalized linear mixed model; [statistical method as in outcome 1, analysis 1]; Count/Rate Ratio = 1.02, 95% CI 2-sided [0.75 to 1.38]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial screening and final follow-up for each participant, a period of approximately 4 months.
Description: We used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | Assessment-only Control | Lab-based Cue Reactivity Personalized Feedback Intervention (PFI)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/51
Other Adverse Events (participants affected / at risk) | 0/42 | 0/51

LIMITATIONS AND CAVEATS:
This is a small pilot trial designed to collect feasibility and acceptability information. The study (enrollment through 3-month) went from May 2023 to March 2024; the COVID-19 pandemic may have impacted alcohol use and contexts of alcohol use. All findings are based on self-report of alcohol use. Analyses reported here restrict the sample to 93 to account for a programming error (subsequently fixed) where control participants were initially being incorrectly emailed a link to the feedback.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT05873556/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT05873556/SAP_001.pdf
  • Informed Consent Form (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT05873556/ICF_002.pdf